CLINICAL TRIAL: NCT04871763
Title: A Protocol for the Assessment of the Bacterial Loads of Essix Retainers in Patients Under Retention Therapy: a Randomized Clinical Trial
Brief Title: Assessment of Bacterial Loads of Essix Retainers in Patients Under Retention Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pavia (Other)
Responsible Party: Principal Investigator, Andrea Scribante, Research Resident, Principal Investigator, University of Pavia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2021-ESSIX
Record Dates: First submitted 2021-04-27; First posted 2021-05-04 (Actual); Last update posted 2021-12-21 (Actual); Status verified 2021-12

CONDITIONS: Orthodontic Appliance Complication
Keywords: oral microbiota; essix retainer; periodontal assessment
MeSH Terms: interventions — Tablets; Water

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Geldis® gel (Experimental): Patients will brush their essix retainers with a toothbrush and with Geldis® gel.
  Interventions: Other: Retainers' Cleansing with Geldis®
- Tablets (Active Comparator): Patients will leave their essix retainers in a glass with water and Polident tablets.
  Interventions: Other: Retainers' Cleansing with tablets
- Water (Active Comparator): Patients will brush essix retainers with a toothbrush under running water.
  Interventions: Other: Retainers' cleansing with water

INTERVENTIONS:
Other: Retainers' Cleansing with Geldis® — Patients will clean their essix retainers with Geldis® using a toothbrush every night for 2 months.
  Arms: Geldis® gel
Other: Retainers' Cleansing with tablets — Patients will leave their essix retainers in a glass with water and Polident tablets every night for 2 months.
  Arms: Tablets
Other: Retainers' cleansing with water — Patients will brush their essix retainers with a toothbrush under water every night for 2 months.
  Arms: Water

SUMMARY:
The aim of this study is to investigate the bacterial loads present on essix retainers in patients' contention therapy. Patients are randomly divided into three groups, depending on the product used for the cleansing of the retainers: Geldis, Polident tablets and water. Microbiological samples were taken from the retainers at the baseline, after 1 and after 2 months, together with Bleeding Index, Plaque Index, BEWE Index and Schiff Air Sensitivity test.

DETAILED DESCRIPTION:
The aim of this study is to investigate the bacterial loads present on essix retainers in patients' contention therapy. Patients who wear essix retainers for contention therapy are randomly divided into three groups, depending on the product used for the cleansing of the retainers: Geldis, Polident tablets and water. Periodontal evaluation and microbiological samples are conducted at the baseline, after 1 and after 2 months.

Bacterial loads are collected from essix retainers, whereas Bleeding Index, Plaque Index, BEWE Index and Schiff Air Sensitivity test are assessed from the patients' mouth.

ELIGIBILITY:
Inclusion Criteria:

* Patients who completed orthodontic treatment and under Essix retainers phase.

Exclusion Criteria:

* Patients under orthodontic treatment with fixed appliances or clear aligners.
* Non-orthodontic patients.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2021-05-12 (Actual); Primary Completion 2021-12-15 (Actual); Study Completion 2021-12-18 (Actual)

PRIMARY OUTCOMES:
Change in PCR% - Plaque Control Record (percentage) | Study begin, 1 and 2 months
  % assessment of the amount of plaque on dental surfaces; it is detected on 4 surfaces: distal, mesial, vestibular, lingual / palatal. The number of sites with plaque is divided by the total number of sites available in the mouth and multiplied by 100. Results indicate the index as a percentage.
Change in BOP - Bleeding on Probing (percentage) | Study begin, 1 and 2 months
  Site-specific assessment of the presence or absence of gum bleeding after the insertion of the periodontal probe for the detection of PPD, detected on 4 sites (mesial, distal, vestibular, palatal/lingual).
  Percentage of sites with bleeding on probing determines the BOP%.
Change in Schiff Air Index - Dental sensitivity test | Study begin, 1 and 2 months
  Scoring criteria:
  * 0: the subject did not respond to air blasting;
  * 1: the subject responded to air blasting;
  * 2: the subject responded to air blasting and requested discontinuation;
  * 3: the subject responded to air blasting, requested discontinuation and considered the stimulus to be painful.
Change of the BEWE Index - Basic Erosive Wear Examination (Barlet et al., 2008) | Study begin, 1 and 2 months
  Scoring criteria:
  0: no erosive tooth wear;
  1. initial loss of surface texture;
  2. distinct defect, hard tissue loss < 50% of the surface area;
  3. hard tissue loss ≥ 50% of the surface area.
Change in microbiological loads of clear aligners | Study begin, 1 and 2 months
  Microbiological assessment of the following loads:
  * Porphyromonas gingivalis
  * Tannarella forsythensis
  * Treponema denticola
  * Peptostreptococcus micros
  * Total bacterial load

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Scribante, DDS, PhD., Principal Investigator — University of Pavia
Locations (1):
- Unit of Dental Hygiene - Section of Dentistry - Department of Clinical, Surgical, Diagnostic and Paediatrics - University of Pavia, Pavia, Lombardy, Italy

IPD SHARING:
Plan to Share IPD: No
Data will be available upon motivated request to Principal Investigator